CLINICAL TRIAL: NCT04753411
Title: Validity and Reliability of The 3-Meter Backward Walk Test in Individuals With Multiple Sclerosis
Brief Title: The 3-Meter Backward Walk Test in Individuals With Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Furkan BİLEK, Lecturer, Firat University
Other Study IDs: Firat U
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Reliability and Validity
Keywords: Multiple Sclerosis; Balance; Backward
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The 3-m backward walk test (3MBWT) is used to evaluate neuromuscular control, proprioception, protective reflexes, fall risk and balance. The aim of our study was to reveal the test-retest reliability and validity of the 3MBWT in Multiple Sclerosis patients.

Our study will be done as a "test-retest" design and psychometric properties of 3 m backward walking test in MS patients will be examined. Mini Mental State Examination, 3 m walk back test, Berg Balance Scale, Timed Up and Go, Timed 25 Step Walking Test and 4-Square Step Test will be applied to the patients. All evaluations will be made by the same physiotherapist. The second and third evaluation (retest) will be performed by the same physiotherapist two days after the first evaluation (test) and 2 weeks later to measure test-retest reliability. It will be preferable to collect data with the same evaluator to avoid inter-rater error rate between evaluations. It will be preferable to collect data with the same evaluator to avoid inter-rater error rate between evaluations.

The sample size, according to Lexell and Downham (2005), 40-50 participants should be included in reliability studies. Considering this recommendation, which defines the reliability of 3MBWT, it is planned to include 50 individuals with MS in our study.

DETAILED DESCRIPTION:
The methodological model of the study is the validity and reliability study. Individuals who applied to Fırat University Training and Research Hospital after ethical approval and diagnosed with MS by a neurologist will be included in our study. It is planned to collect data from individuals who meet the inclusion criteria on a voluntary basis with the Helsinki Declaration. As demographic characteristics; Patients' age, gender, body weight, height, EDSS score, occupation and education status, as a history of the disease, the number of falls in the last year and the type of MS will be recorded. Inclusion criteria for the volunteers; Individuals with relapsing-remitting MS, with an EDSS score between 05≤ and ≤5.5, with an EDSS score between 18-65, and individuals with a score of 24 and above in the Mini Mental State Examination and who can independently walk a minimum of 10 m will be included. Also exclusion criteria for volunteers; High level spasticity of the lower limbs (Ashworth score 3 or 4), who had an acute MS attack or had a history of an attack within the last 1 month, had orthopedic or systemic problems that prevented participation in tests, had another known neuromuscular disorder other than MS, had visual involvement or diplopia, and Having a cardio-pulmonary problem that will prevent him from participating in tests.

Our study will be done as a "test-retest" design and psychometric properties of 3 m backward walking test in MS patients will be examined. Mini Mental State Examination, 3 m walk back test, Berg Balance Scale, Timed Up and Go, Timed 25 Step Walking Test and 4-Square Step Test will be applied to the patients. All evaluations will be made by the same physiotherapist. The second and third evaluation (retest) will be performed by the same physiotherapist two days after the first evaluation (test) and 2 weeks later to measure test-retest reliability. It will be preferable to collect data with the same evaluator to avoid inter-rater error rate between evaluations.

The sample size, according to Lexell and Downham, 30-50 participants should be included in reliability studies . Considering this recommendation, which defines the reliability of 3MBWT, it is planned to include 50 individuals with MS in our study.

Statistical analysis SPSS for Windows 20.00 computer package program will be used for all statistical analyzes. Descriptive statistical information will be given as mean ± standard deviation (x ± SD) or%. Interclass Correlation Coefficients (ICC) and Cronbach's coefficients values will be examined for the reliability and internal consistency of 3MGDYT. The data will be analyzed with appropriate statistical methods and the statistical significance level will be accepted as p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with relapsing-remitting MS, with an EDSS score between 05≤ and ≤5.5, with an EDSS score between 18-65, and individuals with a score of 24 and above in the Mini Mental State Examination and who can independently walk a minimum of 10 m will be included.

Exclusion Criteria:

* Exclusion criteria for volunteers; High level spasticity of the lower limbs (Ashworth score 3 or 4), who had an acute MS attack or had a history of an attack within the last 1 month, had orthopedic or systemic problems that prevented participation in tests, had another known neuromuscular disorder other than MS, had visual involvement or diplopia, and Having a cardio-pulmonary problem that will prevent him from participating in tests.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals who applied to Fırat University Training and Research Hospital and diagnosed with MS by a neurologist will be included.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-02-05 (Estimated); Primary Completion 2021-04-04 (Estimated); Study Completion 2021-05-04 (Estimated)

PRIMARY OUTCOMES:
3 Meter Backward Walking Test | 2 weeks
  The 3-meter distance is marked with a black tape and the participants are asked to align their heels with black tape. Individuals are asked to walk backwards as soon as possible with the "walk" command and stop when they reach 3 meters. Meanwhile, the elapsed time is recorded in seconds. The evaluation will take place three times and the average time will be recorded.
Berg Balance Scale | 1 day
  It was designed for quantitative evaluation of balance and determination of fall risk, and was chosen because it evaluates individuals' ability to maintain their balance while performing functional activities. According to the scores obtained from the test in question, the cases were divided into groups as "high fall risk (0-20 points)", "medium fall risk (21-40 points)", "low fall risk (41-56)". score) ". Fifty-six, the highest score, is considered to show the best balance. Turkish validity and reliability study of the scale was conducted by Şahin et al.
Timed Get Up and Go Test | 1 day
  It is applied to assess the balance and fall risk of individuals. The patient is first asked to sit on a chair. The patient is then asked to stand up, walk regularly at a predetermined distance of 3 meters, return at the end of 3 meters and sit on a chair. The walking time of the patient during the test is recorded with the stopwatch in seconds. The test was repeated three times and the average value will be recorded
4-Square Step Test | 1 day
  Aims to evaluate dynamic balance and stepping forward, side and back over objects. Using tape, 1 horizontal and 1 vertical line is made in the form of diagonal 4 divisions. At the start of the test, the individual stands in the upper left square. Then they step clockwise with both feet before moving on to the next frame: first to the right, then back, then to the left, and finally to the back position. They immediately follow this by stepping counterclockwise. After 1 application attempt, the time is saved for the next 2 attempts and the best 1 attempt is counted. Among older adults living in the community, over 15 seconds has been associated with an increased risk of falling

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Frohman EM, Racke MK, Raine CS. Multiple sclerosis--the plaque and its pathogenesis. N Engl J Med. 2006 Mar 2;354(9):942-55. doi: 10.1056/NEJMra052130. No abstract available. PMID 16510748
- [Background] Pelfrey CM, Cotleur AC, Lee JC, Rudick RA. Sex differences in cytokine responses to myelin peptides in multiple sclerosis. J Neuroimmunol. 2002 Sep;130(1-2):211-23. doi: 10.1016/s0165-5728(02)00224-2. PMID 12225904
- [Background] Frzovic D, Morris ME, Vowels L. Clinical tests of standing balance: performance of persons with multiple sclerosis. Arch Phys Med Rehabil. 2000 Feb;81(2):215-21. doi: 10.1016/s0003-9993(00)90144-8. PMID 10668778
- [Background] Williams NP, Roland PS, Yellin W. Vestibular evaluation in patients with early multiple sclerosis. Am J Otol. 1997 Jan;18(1):93-100. PMID 8989958
- [Background] Daley ML, Swank RL. Quantitative posturography: use in multiple sclerosis. IEEE Trans Biomed Eng. 1981 Sep;28(9):668-71. doi: 10.1109/TBME.1981.324761. No abstract available. PMID 7319527
- [Background] Lanzetta D, Cattaneo D, Pellegatta D, Cardini R. Trunk control in unstable sitting posture during functional activities in healthy subjects and patients with multiple sclerosis. Arch Phys Med Rehabil. 2004 Feb;85(2):279-83. doi: 10.1016/j.apmr.2003.05.004. PMID 14966714
- [Background] Cattaneo D, De Nuzzo C, Fascia T, Macalli M, Pisoni I, Cardini R. Risks of falls in subjects with multiple sclerosis. Arch Phys Med Rehabil. 2002 Jun;83(6):864-7. doi: 10.1053/apmr.2002.32825. PMID 12048669
- [Background] DeBolt LS, McCubbin JA. The effects of home-based resistance exercise on balance, power, and mobility in adults with multiple sclerosis. Arch Phys Med Rehabil. 2004 Feb;85(2):290-7. doi: 10.1016/j.apmr.2003.06.003. PMID 14966716
- [Background] Hobart JC, Riazi A, Lamping DL, Fitzpatrick R, Thompson AJ. Measuring the impact of MS on walking ability: the 12-Item MS Walking Scale (MSWS-12). Neurology. 2003 Jan 14;60(1):31-6. doi: 10.1212/wnl.60.1.31. PMID 12525714
- [Background] Tesio L, Perucca L, Franchignoni FP, Battaglia MA. A short measure of balance in multiple sclerosis: validation through Rasch analysis. Funct Neurol. 1997 Sep-Oct;12(5):255-65. PMID 9439943
- [Background] Thomas MA, Fast A. One step forward and two steps back: the dangers of walking backwards in therapy. Am J Phys Med Rehabil. 2000 Sep-Oct;79(5):459-61. doi: 10.1097/00002060-200009000-00011. PMID 10994888
- [Background] Carter V, Jain T, James J, Cornwall M, Aldrich A, de Heer HD. The 3-m Backwards Walk and Retrospective Falls: Diagnostic Accuracy of a Novel Clinical Measure. J Geriatr Phys Ther. 2019 Oct/Dec;42(4):249-255. doi: 10.1519/JPT.0000000000000149. PMID 29095771
- [Background] Rose DK, DeMark L, Fox EJ, Clark DJ, Wludyka P. A Backward Walking Training Program to Improve Balance and Mobility in Acute Stroke: A Pilot Randomized Controlled Trial. J Neurol Phys Ther. 2018 Jan;42(1):12-21. doi: 10.1097/NPT.0000000000000210. PMID 29232308
- [Background] Abit Kocaman A, Aydogan Arslan S, Ugurlu K, Katirci Kirmaci ZI, Keskin ED. Validity and Reliability of The 3-Meter Backward Walk Test in Individuals with Stroke. J Stroke Cerebrovasc Dis. 2021 Jan;30(1):105462. doi: 10.1016/j.jstrokecerebrovasdis.2020.105462. Epub 2020 Nov 13. PMID 33197801
- [Background] Lexell JE, Downham DY. How to assess the reliability of measurements in rehabilitation. Am J Phys Med Rehabil. 2005 Sep;84(9):719-23. doi: 10.1097/01.phm.0000176452.17771.20. PMID 16141752
- [Background] Sahin F, Yilmaz F, Ozmaden A, Kotevolu N, Sahin T, Kuran B. Reliability and validity of the Turkish version of the Berg Balance Scale. J Geriatr Phys Ther. 2008;31(1):32-7. doi: 10.1519/00139143-200831010-00006. PMID 18489806
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Roos MA, Reisman DS, Hicks G, Rose W, Rudolph KS. Development of the Modified Four Square Step Test and its reliability and validity in people with stroke. J Rehabil Res Dev. 2016;53(3):403-12. doi: 10.1682/JRRD.2014.04.0112. PMID 27271003